CLINICAL TRIAL: NCT06367894
Title: Study on Treatment Optimization and Nephrolithiasis Recurrence Prevention With Interdisciplinary Care
Brief Title: Treatment Optimization and Nephrolithiasis Recurrence Prevention With Interdisciplinary Care
Status: Recruiting | Type: Observational
Sponsor: Agnieszka Pozdzik (Other)
Responsible Party: Sponsor-Investigator, Agnieszka Pozdzik, Head of nephrology clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: STONECARE
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nearly 10% of the Belgian population suffer from kidney stone disease. Recent reviews reported that kidney stones represent an underestimated risk factor for further kidney function deterioration. Preventive measures are recommended in lithiases patients to prevent the formation of new stones. The individual effects of different medicated prosthetic interventions have been documented in clinical trials. However, there is little data on the effectiveness of combining these different preventive measures in routine clinical practice (real-world context).

Patients with kidney stone disease require a complete metabolic assessment. The three main factors contributing to the stone's formation are the patient's metabolism, diet and lifestyle. Metabolic work-up is recommended by the American Urology Association to identify and correct the factors responsible for urinary stone formation such as hypercalciuria, hyperoxaluria, hyperuricuria, hypocitraturia or abnormalities of urinary pH. The metabolic work-up includes at minimum the 24h urine test, a blood test and spot urine test. Dietary habits and lifestyle are assessed by means of a questionnaire.

The CHU Brugmann Hospital has a specialized multidisciplinary clinic for renal lithiases and mineral metabolism. Preventive personalized and interdisciplinary care in CHU Brugmann consists of a full metabolic work-up allowing the identification of lithogenic risk factors by nephrologists, dietary assessment by specialized dieticians and specific treatment protocol associated with regular follow-up.

The aim of this study is to evaluate, in the context of a retrospective single-center cohort study, the effect of preventive personalized and interdisciplinary care on the evolution of all urinary lithogenic risk factors and the recurrence of kidney stones (rate of renal colics, emergency room admissions, and urological interventions).

ELIGIBILITY:
Inclusion Criteria:

* All patients of the CHU Brugmann Hospital who fulfill the criteria of active or past history of kidney stone, from 01/01/2018 till 31/10/2023
* Minimum follow-up time of 2 months with biochemical and clinical results available

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of the CHU Brugmann Hospital who fulfill the criteria of active or past history of kidney stone, from 01/01/2018 till 31/10/2023
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of acute renal colics | From first patient consultation till 31/10/2023
  Number of acute renal colics
Number of emergency admissions | From first patient consultation till 31/10/2023
  Number of emergency admissions
Number of surgeries | From first patient consultation till 31/10/2023
  Number of surgeries
Number of hospitalizations | From first patient consultation till 31/10/2023
  Number of hospitalizations
Identified genetics abnormalities | From first patient consultation till 31/10/2023
  List of identified genetics abnormalities
Wisconsin questionnaire | From first patient consultation till 31/10/2023
  Changes in the quality of life in the patients (evolution of the scoring of the Wisconsin questionnaire)
Kidney function outcome | Status at 31/10/2023
  Kidney function outcome

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No